CLINICAL TRIAL: NCT00005689
Title: Trial of Smoking Cessation Programs in Black Churches
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4185
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Heart Disease Risk Reduction
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
To provide a comprehensive description of smoking beliefs and behavior among rural Blacks, and to test the effectiveness of smoking cessation strategies delivered through Black churches.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

Two demographically similar rural counties in central Virginia were compared, one intervention and one control site. In each country, two cohorts were assembled, a random sample of all Black smokers (the community cohort), and all members of randomly sampled Black churches (the church cohort). The descriptive component of the study elicited the knowledge, beliefs, attitudes, and behavior concerning smoking from these cohorts. Cardiovascular risk factors, including blood pressure and cholesterol levels, were also determined in the community cohort. For the experimental component, a variety of interventions which have proven to be efficacious in other settings were implemented through Black churches. These included fostering a supportive environment, distributing self-help materials, and providing individual support and counselling through the use of peer facilitators. The results of the baseline psychosocial survey were used to modify these methods for local use. They were then implemented in a culturally appropriate fashion at the intervention sites. Baseline smoking rates were determined using the initial surveys in both counties. Smokers were surveyed again at the end of the interventions and one year later to establish one-year abstinence rates. These were used as the primary outcome variables for the analysis of effect. The principal effect of the interventions were measured by comparing smoking abstinence rates between the church cohorts in the intervention and control counties. Due to the extended nature of the social networks associated with the churches, the interventions may also have had an effect on individuals not directly exposed, and this was determined by comparing the outcomes in the community cohorts. Finally, the associations between the baseline psychosocial and physiologic variables, exposure to the interventions, and smoking cessation behavior were also analyzed, to characterize on a population basis those who were and were not influenced by these church-based programs.

ELIGIBILITY:
No eligibility criteria

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-07; Study Completion 1995-06

REFERENCES:
- [Background] Willems JP, Saunders JT, Hunt DE, Schorling JB. Prevalence of coronary heart disease risk factors among rural blacks: a community-based study. South Med J. 1997 Aug;90(8):814-20. doi: 10.1097/00007611-199708000-00008. PMID 9258308
- [Background] Schorling JB, Roach J, Siegel M, Baturka N, Hunt DE, Guterbock TM, Stewart HL. A trial of church-based smoking cessation interventions for rural African Americans. Prev Med. 1997 Jan-Feb;26(1):92-101. doi: 10.1006/pmed.1996.9988. PMID 9010903
- [Background] Willems JP, Hunt DE, Schorling JB. Coronary heart disease risk factors and cigarette smoking among rural African Americans. J Natl Med Assoc. 1997 Jan;89(1):37-47. PMID 9002415
- [Background] Schorling JB. The stages of change of rural African-American smokers. Am J Prev Med. 1995 May-Jun;11(3):170-7. PMID 7662396